CLINICAL TRIAL: NCT02316067
Title: Effect of Corporal Suspension and Pendulum Exercises on Torque, Muscle Activation, Muscle Thickness and Functionality in Patients With Traumatic Spinal Cord Injury
Brief Title: Traumatic Spinal Cord Injury: Effects of Corporal Suspension and Pendulum Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marco Aurélio Vaz, PhD (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor-Investigator, Marco Aurélio Vaz, PhD, PhD, Federal University of Rio Grande do Sul
Organization: Federal University of Rio Grande do Sul (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UFRGS - 70254
Record Dates: First submitted 2014-12-08; First posted 2014-12-12 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal cord; Wounds and Injuries; Rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries; Wounds and Injuries | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rehabilitation (Experimental): Eight weeks of rehabilitation (CHORDATA® Method)
  Interventions: Other: Rehabilitation
- Control (No Intervention): Participants maintained their daily-life activities routine during the same eight weeks period and were tested before and after this control period.

INTERVENTIONS:
Other: Rehabilitation — The CHORDATA® Method (16 sessions; 50 minutes each; twice a week) consisted of three exercises: (1) anterior pendulum, with the patient seated on a chair, upper limb suspended by springs and straps, and actively moving the trunk forward; (2) posterior pendulum exercise, on a similar position as exercise (1) but now moving the trunk backwards and recruiting the abdominal wall muscles during a posterior pelvic tilt motion; and (3) stand-up and sit-down exercise, patient with knees fixed anteriorly, initiating the standing-up movement by pulling back and down the springs, trying to maintain the standing position for as long as possible, balancing the trunk and transferring the supporting force from the upper limbs to the lower limbs.
  Arms: Rehabilitation

SUMMARY:
The purpose of this study was to evaluate the effects of an exercise program proposed by the CHORDATA® Method on the functionality, maximal isometric torque, muscle activity and muscle thickness of trunk muscles in patients with traumatic spinal cord injury.

The hypothesis is that the CHORDATA® Method could reduce the deleterious effects of the traumatic spinal cord injury.

DETAILED DESCRIPTION:
Participants were allocated into one of two groups (rehabilitation or control). Rehabilitation group (8 weeks of rehabilitation; CHORDATA® Method) Control group (patients with up to three years of traumatic spinal cord injury): Participants maintained their daily-life activities routine during the same eight weeks period and were tested before and after this control period. At the end of the control period, patients interested at participating on the training program were included in the intervention group

ELIGIBILITY:
Inclusion Criteria:

- Patients that suffered traumatic spinal cord injury in the last 42 months, capable of transporting themselves for rehabilitation at the physical therapy clinic and for the neuromuscular tests at the laboratory where measurements were performed.

Exclusion Criteria:

* Body weight above 95kg
* Physical and functional limitations impeding them of performing physical activity
* Physically incapacitating diseases (e.g severe cardiovascular and respiratory diseases, neurodegenerative diseases, oncologic diseases, systemic arterial hypertension)
* Visual deficit that impeded reading
* Recurrent vertigo or hypotension to exercise
* Engaged in other treatments that could constitute a confounding effect
* Changed their daily life activities during the study

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-05; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Torque change ( assessed by dynamometry.) | Torque was measured 2 times during the study: Pre-intervention/control and post-intervention/control (8 weeks after the first assessment).
  Torque is an expression of the muscular strength and was assessed by dynamometry.

SECONDARY OUTCOMES:
Muscular electrical activation change (assessed by electromyography (EMG) | Muscular electrical activation was measured 2 times during the study: Pre-intervention/control and post-intervention/control (8 weeks after the first assessment).
  Electrical activation was assessed by electromyography (EMG).

OTHER OUTCOMES:
Muscle thickness change (assessed by ultrasonography) | Muscle thickness was measured 2 times during the study: Pre-intervention/control and post-intervention/control (8 weeks after the first assessment).
  Muscle thickness was assessed by ultrasonography
Functional performance change (assessed by Functional Reach Adapted Test) | Functional performace was measured 2 times during the study: Pre-intervention/control and post-intervention/control (8 weeks after the first assessment).
  Functional performance was assessed by Functional Reach Adapted Test

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Netto, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Exercise Research Laboratory, School of Physical Education, Federal University of Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Frison VB, Lanferdini FJ, Geremia JM, de Oliveira CB, Radaelli R, Netto CA, Franco AR, Vaz MA. Effect of corporal suspension and pendulum exercises on neuromuscular properties and functionality in patients with medullar thoracic injury. Clin Biomech (Bristol). 2019 Mar;63:214-220. doi: 10.1016/j.clinbiomech.2019.02.012. Epub 2019 Feb 23. PMID 30952032